CLINICAL TRIAL: NCT01859923
Title: Phase 2, Open-label, Multiple-dose Trial to Assess the Safety, Tolerability, Pharmacokinetics, and Efficacy of Delamanid (OPC-67683) in Pediatric Multidrug-resistant Tuberculosis Patients on Therapy With an Optimized Background Regimen of Anti-tuberculosis Drugs Over a 6-Month Treatment Period
Brief Title: A 6-Month Safety, Efficacy, and Pharmacokinetic (PK) Trial of Delamanid in Pediatric Participants With Multidrug Resistant Tuberculosis (MDR-TB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 242-12-233; 2012-004620-38 (EudraCT Number)
Record Dates: First submitted 2013-05-15; First posted 2013-05-22 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Multidrug Resistant Tuberculosis
Keywords: Tuberculosis; Tuberculosis, Multidrug-Resistant; Mycobacterium Infections; Actinomycetes Infections; Gram-Positive Infections; Bacterial Infections; Pediatric
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Tuberculosis; Mycobacterium Infections; Bacterial Infections | interventions — OPC-67683

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: 12 to 17 Years of Age (Experimental): Participants 12 to 17 years old (inclusive) received adult formulation of delamanid 100 milligrams (mg) (2x50 mg tablets), orally, twice daily (BID) plus optimized background regimen (OBR) up to Day 182. Participants continued to receive OBR up to Day 365.
  Interventions: Drug: Delamanid; Drug: Optimized Background Regimen (OBR)
- Group 2: 6 to 11 Years of Age (Experimental): Participants 6 to 11 years old (inclusive) received adult formulation delamanid 50 mg (1x50 mg tablet), orally, BID plus OBR up to Day 182. Participants continued to receive OBR up to Day 365.
  Interventions: Drug: Delamanid; Drug: Optimized Background Regimen (OBR)
- Group 3: 3 to 5 Years of Age (Experimental): Participants 3 to 5 years old (inclusive) received 25 mg pediatric formulation of delamanid (DPF - suspension prepared using dispersible tablet), orally, BID plus OBR up to Day 182. Participants continued to receive OBR up to Day 365.
  Interventions: Drug: Delamanid Pediatric Formulation (DPF); Drug: Optimized Background Regimen (OBR)
- Group 4: Birth to 2 Years of Age (Experimental): Participants from birth to 2 years old (inclusive) received DPF (suspension prepared using dispersible tablet) for 182 days plus OBR. Participants continued to receive OBR up to Day 365. The DPF dose was based on the participant's body weight during the baseline visit:
  * Participants >10 kilograms (kg) received DPF 10 mg BID plus OBR
  * Participants >8 kg and ≤10 kg received DPF 5 mg BID plus OBR
  * Participants ≥5.5 kg and ≤8 kg received DPF 5 mg once per day (QD) plus OBR
  Delamanid dose was adjusted as needed for Group 4 participants based on the weight measurement at specified study visits [Visits 5 (Day 28), 7 (Day 56), 9 (Day 84), 11 (Day 126) and 12 (Day 154)].
  Interventions: Drug: Delamanid Pediatric Formulation (DPF); Drug: Optimized Background Regimen (OBR)

INTERVENTIONS:
Drug: Delamanid — Participants received adult formulation delamanid as per regimen specified in the arm description. Morning dose of the delamanid BID regimen was given within 30 minutes after the start of a standard breakfast meal. The evening dose of the BID dose regimen was given 10 hours post morning dose and within 30 minutes after the start of a standard dinner meal.
  Other Names: OPC-67683
  Arms: Group 1: 12 to 17 Years of Age; Group 2: 6 to 11 Years of Age
Drug: Delamanid Pediatric Formulation (DPF) — Participants received delamanid as an extemporaneous suspension using the delamanid pediatric dispersible tablet formulation. Morning dose of the delamanid BID/once daily (QD) regimen was given within 30 minutes after the start of a standard breakfast meal. The evening dose of the BID dose regimen was given 10 hours post morning dose and within 30 minutes after the start of a standard meal.
  Arms: Group 3: 3 to 5 Years of Age; Group 4: Birth to 2 Years of Age
Drug: Optimized Background Regimen (OBR) — Selection and administration of the treatment medications (i.e. OBRs) was based on Search Results Web result with site links
  World Health Organization (WHO's) Guidelines for the programmatic management of drug-resistant TB, in conjunction with national TB program guidelines. Study Investigator could change OBR for a participant based on his/her tolerability and drug susceptibility testing (DST) results.

SUMMARY:
The purpose of this trial is to assess the safety, tolerability, pharmacokinetics, and efficacy of long-term (6-month) treatment with delamanid plus an optimized background regimen (OBR) of other anti-tuberculosis drugs in pediatric participants who completed Study 242-12-232 (NCT01856634).

DETAILED DESCRIPTION:
This study will assess the safety, tolerability, pharmacokinetics, and efficacy of delamanid plus an optimized background regimen in pediatric participants with MDR-TB over a 6-month treatment period. This long-term study, an extension of Study 242-12-232, will be conducted in participants who have completed Study 242-12-232.

ELIGIBILITY:
Inclusion Criteria:

* Successfully completed Trial 242-12-232
* Confirmed diagnosis of MDR-TB OR
* Presumptive diagnosis of pulmonary or extrapulmonary MDR-TB including one of the following:

  * Clinical specimen suggestive of tuberculosis disease
  * Persistent cough lasting > 2 weeks
  * Fever, weight loss, and failure to thrive
  * Findings on recent chest radiograph (prior to Visit 1) consistent with TB AND
  * Household contact with a person with known MDR-TB or with a person who died while appropriately taking drugs for sensitive TB OR
  * On first-line TB treatment but with no clinical improvement
* Negative urine pregnancy test for female participants who have reached menarche
* Written informed consent/assent

Exclusion Criteria:

* Participants who have not completed Trial 242-12-232
* Laboratory evidence of active hepatitis B or C
* Children with body weight < 5.5 kg
* For participants with human-immunodeficiency virus (HIV) co-infection, cluster difference-4 (CD4) cell count ≤ 1000/mm^3 for children 1-5 years old, and ≤ 1500/mm^3 for children less than 1 year old
* History of allergy to metronidazole and any disease or condition in which metronidazole is required
* Use of amiodarone within 12 months or use of other predefined antiarrhythmic medications within 30 days prior to first dose of delamanid
* Serious concomitant conditions
* Pre-existing cardiac conditions
* Abnormalities in Screening electrocardiogram (ECG) [including atrio-ventricular (AV) block, blood brain barrier (BBB) or hemi-block, QRS prolongation > 120 milliseconds (ms), or QT interval corrected by Fridericia's formula (QTcF) > 450 ms in both males and females]
* Concomitant condition such as renal impairment characterized by serum creatinine levels > 1.5 mg/dL, hepatic impairment (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3x upper limit of normal (ULN)), or hyperbilirubinemia characterized by total bilirubin > 2x ULN
* Current diagnosis of severe malnutrition or kwashiorkor
* Positive urine drug screen (Groups 1 and 2 only)
* Rifampicin and/or moxifloxacin within 1 week prior to the first dose of delamanid and/or any prior or concurrent use of bedaquiline
* Lansky Play Performance Score < 50 (not applicable for children < 1 year old) or Karnofsky Score < 50
* Administered an investigational medicinal product (IMP) within 1 month prior to Visit 1 other than delamanid given as IMP in Trial 242-12-232
* Pregnant, breast-feeding, or planning to conceive or father a child within the timeframe described in the informed consent form (Groups 1 and 2 only)

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2013-07-20 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melchor VG Frias, IV, MD, Principal Investigator — De La Salle Health Sciences Institute; Anjanette Reyes-De Leon, MD, Principal Investigator — Lung Center of the Philippines; Louvina van der Laan, MD, Principal Investigator — Brooklyn Chest Hospital
Locations (3):
- Philippines (2):
  - De La Salle Health Sciences Institute, Dasmariñas, Cavite
  - Lung Center of the Philippines, Quezon City, National Capital Region
- Brooklyn Chest Hospital, Ysterplaat, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Garcia-Prats AJ, Frias M, van der Laan L, De Leon A, Gler MT, Schaaf HS, Hesseling AC, Malikaarjun S, Hafkin J. Delamanid Added to an Optimized Background Regimen in Children with Multidrug-Resistant Tuberculosis: Results of a Phase I/II Clinical Trial. Antimicrob Agents Chemother. 2022 May 17;66(5):e0214421. doi: 10.1128/aac.02144-21. Epub 2022 Apr 11. PMID 35404075

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in study at 3 investigative sites in Philippines and South Africa from July 20, 2013 to January 13, 2020. Participants received delamanid up to Day 182 in the treatment period and were followed up to Day 365 for safety and efficacy and up to Day 730 (Month 24) for treatment outcome.
Pre-assignment Details: Pediatric participants with a diagnosis of multidrug-resistant tuberculosis (MDR-TB) who were on therapy with an optimized background regimen (OBR) of anti-tuberculosis drugs and completed study 242-12-232 (NCT01856634) were enrolled in this extension study 242-12-233 to receive delamanid based on the participant's age and weight.
Period: Overall Study
Arm/Group | Group 1: 12 to 17 Years of Age | Group 2: 6 to 11 Years of Age | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age
Started | 7 | 6 | 12 | 12
Completed | 7 | 6 | 11 | 11
Not Completed | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Sample included participants who received any amount of investigational medicinal product (IMP) in this study, regardless of any protocol deviation or violation.
Groups:
- Group 1: 12 to 17 Years of Age: Participants 12 to 17 years old (inclusive) received adult formulation of delamanid 100 mg (2x50 mg tablets), orally, BID plus OBR up to Day 182. Participants continued to receive OBR up to Day 365.
- Total: Total of all reporting groups
Arm/Group | Group 1: 12 to 17 Years of Age | Group 2: 6 to 11 Years of Age | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age | Total
Number analyzed (Participants) | 7 | 6 | 12 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.37 (1.63) | 9.51 (1.49) | 4.37 (0.98) | 1.79 (0.59) | 6.45 (5.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 6 | 6 | 19
  Male | 4 | 2 | 6 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 12 | 12 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 2 | 0 | 2
  Asian | 7 | 4 | 8 | 6 | 25
  Other | 0 | 2 | 2 | 6 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  Philippines | 7 | 4 | 8 | 6 | 25
  South Africa | 0 | 2 | 4 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With At Least One Treatment Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant and that does not necessarily have a causal relationship with the treatment. A TEAE is defined as an AE that occurred after the administration of investigational medicinal product (IMP).
Time Frame: From the first dose of study drug up to the end of the Post-treatment Follow-up Period (Up to Day 365)
Population: The Safety Sample included participants who received any amount of IMP in this study, regardless of any protocol deviation or violation.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 12 to 17 Years of Age | Group 2: 6 to 11 Years of Age | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age
Number analyzed (Participants) | 7 | 6 | 12 | 12
Participants | 7 | 6 | 12 | 12

2. Primary Outcome: Number of Participants With Abnormal Physical Examination Values
Description: Physical examination included the examination of the abdomen; extremities; head, eyes, ears, nose (HEENT); neurological; skin and mucosae; thorax; urogenital; audiometry assessment and visual assessment. Participants with abnormal values, as assessed by the investigator were reported.
Time Frame: From the first dose of study drug up to the end of the Post-treatment Follow-up Period (Up to Day 365)
Population: The Safety Sample included participants who received any amount of IMP in this study, regardless of any protocol deviation or violation. Overall number of participants analyzed are the participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 12 to 17 Years of Age | Group 2: 6 to 11 Years of Age | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age
Number analyzed (Participants) | 7 | 6 | 12 | 11
Participants
  Abdomen | 1 | 1 | 4 | 2
  Extremities | 2 | 0 | 1 | 1
  HEENT | 7 | 6 | 12 | 10
  Neurological | 1 | 0 | 1 | 1
  Skin and Mucosae | 2 | 6 | 6 | 8
  Thorax | 5 | 2 | 6 | 7
  Urogenital | 0 | 0 | 1 | 3
  Audiometry Assessment | 4 | 3 | 9 | 7
  Visual Assessment | 0 | 1 | 0 | 1

3. Primary Outcome: Number of Participants With Clinically Significant Abnormal Vital Sign Values
Description: Vital signs included weight (kg), height (cm), body temperature (degree Celsius), heart rate (beats/min), respiratory rate (breaths/minute), systolic and diastolic blood pressure (mm Hg), body mass index (BMI) (kg/m^2). The criteria for clinically significant abnormal value for weight was decrease or increase of >=5% in body weight relative to Baseline. Only categories with data for potentially clinically significant abnormal vital sign parameter values are reported.
Time Frame: From the first dose of study drug up to the end of the Post-treatment Follow-up Period (Up to Day 365)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 12 to 17 Years of Age | Group 2: 6 to 11 Years of Age | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age
Number analyzed (Participants) | 7 | 6 | 12 | 11
Participants
  Decrease of >=5% in Body Weight | 0 | 2 | 0 | 1
  Increase of >=5% in Body Weight | 4 | 2 | 10 | 10

4. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) Values
Description: The criteria for clinically significant abnormal ECG values were ventricular rate outlier (<50 bpm and decrease of >=25%, >100 bpm and increase of >=25%), PR outlier (increase of >=25% when PR >200 milliseconds (ms)), QRS outlier (increase of >=25% when QRS >100 ms), QT (new onset (in treatment period but not at Baseline) [>500 ms]), QT interval corrected by Bazett's formula (QTcB) (new onset [>450, >480, >500 ms], increase of >=30 ms and <= 60 ms or increase of >60 ms), QT interval corrected by Fridericia's formula (QTcF) (new onset [>450, >480, >500 ms], increase of >=30 ms and <= 60 ms or increase of >60 ms), new abnormal U waves, new ST segment changes, new T wave changes, new abnormal rhythm, new conduction abnormality were reported as categories. Only categories with data are reported.
Time Frame: From the first dose of study drug up to the end of the Post-treatment Follow-up Period (Up to Day 365)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 12 to 17 Years of Age | Group 2: 6 to 11 Years of Age | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age
Number analyzed (Participants) | 7 | 6 | 12 | 11
Participants
  Ventricular Rate Outliers, Notable Increases | 1 | 0 | 1 | 4
  QRS Outliers | 1 | 0 | 0 | 0
  QTcB, New Onset (>480 ms) | 1 | 1 | 1 | 0
  QTcB, New Onset (>450 ms) | 7 | 2 | 8 | 5
  QTcB, New Onset (Change >= 30 and <=60 ms) | 5 | 3 | 8 | 9
  QTcB, New Onset (Change > 60 ms) | 1 | 0 | 0 | 2
  QTcF, New Onset (>450 ms) | 3 | 2 | 0 | 0
  QTcF, New Onset (Change >= 30 and <=60 ms) | 5 | 2 | 6 | 9
  QTcF, New Onset (Change > 60 ms) | 1 | 0 | 0 | 1
  New Abnormal Rhythm | 5 | 4 | 6 | 1
  New Conduction Abnormality | 6 | 5 | 5 | 8

5. Primary Outcome: Number of Participants With Clinically Significant Laboratory Test Abnormalities
Description: Laboratory assessments included parameters for serum chemistry, hematology and urinalysis along with adrenocorticotropic hormone, serum cortisol, free thyroxine, thyroid-stimulating hormone (TSH), and high sensitivity C-reactive protein cell count. The participants were categorized based on the clinically significant laboratory values as per protocol predefined criteria. The categories with at least one participant with clinically significant value outside the normal range for laboratory assessments are reported. The normal ranges for those laboratory parameters were potassium 3.4 - 5.4 milliequivalents/liter (mEq/L), uric acid 3.9 - 8.2 mg/dL, partial thromboplastin time (PTT) 9.7 - 12.3 sec, platelet count 180 - 440 thousands platelets/μL.
Time Frame: From the first dose of study drug up to the end of the Post-treatment Follow-up Period (Up to Day 365)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 12 to 17 Years of Age | Group 2: 6 to 11 Years of Age | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age
Number analyzed (Participants) | 7 | 6 | 12 | 12
Participants
  Elevated Potassium | 0 | 0 | 0 | 1
  Elevated Uric Acid | 1 | 0 | 1 | 0
  Elevated PTT | 0 | 1 | 2 | 0
  Low Platelet Count | 0 | 0 | 0 | 1

6. Primary Outcome: Population Pharmacokinetic (POPPK) Model Point Estimate for Central Clearance (L) and Inter-compartmental Clearance (Q) of Delamanid
Description: Central clearance is defined as plasma volume in the vascular compartment that is cleared of drug per unit of time. Inter-compartmental clearance is defined as a ratio of the drug's distribution rate between the central compartment and the peripheral compartments over its circulating concentration (L/hr). Population point estimates were based on POPPK analysis to find one measure each for both L and Q. The exposure data were pooled across visits and participants to identify POPPK parameter estimates and were reported for delamanid.
Time Frame: Predose on Days 1, 56, 154, and 182, 210 and at any time point on Days 14, 98, 189, 196, 203, and 238
Population: Population Pharmacokinetic (PK)/Pharmacodynamic (PD) analysis sample included all the participants with data available for PK/PD analysis.
Measure: Number; unit: L/hr
Groups:
- Delamanid: Participants received delamanid 25, 50 or 100 mg based on age and weight plus OBR up to Day 182. Participants continued to receive OBR up to Day 365.
Arm/Group | Delamanid
Number analyzed (Participants) | 37
L/hr
  Central Clearance (L) | 18.1
  Inter-compartmental Clearance (Q) | 105

7. Primary Outcome: POPPK Model Point Estimate for Central Volume of Distribution (Vc) and Peripheral Volume of Distribution (Vp) of Delamanid
Description: Vc is defined as the theoretical volume that would be necessary to contain the total amount of an administered drug at the same concentration that it is observed in the blood plasma. Vp is defined as the apparent volume needed to account for the total amount of drug in the body if the drug was evenly distributed throughout the body and in the same concentration as the site of sample collection such as peripheral venous plasma. Population point estimates were based on POPPK analysis to find one measure each for both Vc and Vp. The exposure data were pooled across visits and participants to identify POPPK parameter estimates and were reported for delamanid.
Time Frame: Predose on Days 1, 56, 154, and 182, 210 and at any time point on Days 14, 98, 189, 196, 203, and 238
Population: Population PK/PD analysis sample included all the participants with data available for PK/PD analysis.
Measure: Number; unit: liters (L)
Arm/Group | Delamanid
Number analyzed (Participants) | 37
liters (L)
  Central Volume of Distribution (Vc) | 254
  Peripheral Volume of Distribution (Vp) | 347

8. Primary Outcome: POPPK Model Point Estimate for Absorption Rate Constant (Ka) of Delamanid
Description: Ka is defined as a measure of rate at which a drug enters into the circulatory system. Population point estimate for Ka was based on population PK analysis to find one measure. Population point estimates were based on POPPK analysis to find one measure for Ka. The exposure data were pooled across visits and participants to identify POPPK parameter estimates and were reported for delamanid.
Time Frame: Predose on Days 1, 56, 154, and 182, 210 and at any time point on Days 14, 98, 189, 196, 203, and 238
Population: Population PK/PD analysis sample included all the participants with data available for PK/PD analysis.
Measure: Number; unit: per hour (1/hr)
Arm/Group | Delamanid
Number analyzed (Participants) | 37
per hour (1/hr) | 0.254

9. Primary Outcome: POPPK Model Point Estimate for Absorption Lag Time (ALAG1) of Delamanid
Description: ALAG1 is defined as the time delay prior to the commencement of drug absorption. Population point estimates were based on POPPK analysis to find one measure for ALAG1. The exposure data were pooled across visits and participants to identify POPPK parameter estimates and were reported for delamanid.
Time Frame: Predose on Days 1, 56, 154, and 182, 210 and at any time point on Days 14, 98, 189, 196, 203, and 238
Population: Population PK/PD analysis sample included all the participants with data available for PK/PD analysis.
Measure: Number; unit: hour (hr)
Arm/Group | Delamanid
Number analyzed (Participants) | 37
hour (hr) | 1.38

10. Secondary Outcome: Baseline QT Interval (QTcB) Effect
Description: The 12-lead ECG was performed to obtain recordings of heart rate (QT interval) to analyze QTcB effect.
Time Frame: Baseline (Day -1)
Population: Population PK/PD analysis sample included all the participants with data available for PK/PD analysis.
Measure: Mean (90% Confidence Interval); unit: ms
Arm/Group | Delamanid
Number analyzed (Participants) | 37
ms
  Delamanid | 0.0318 [-0.113 to 0.177]
  Metabolite DM-6705 | 0.0309 [-0.112 to 0.174]

11. Secondary Outcome: PK/PD Relationship: POPPK Model Point Estimate for Slope of Linear Mixed Effects Model for Change in QTcB Interval Versus Delamanid Plasma Concentrations
Description: The linear mixed effects model was applied to characterize the concentration-QTcB relationship of delamanid/DM-6705 to obtain population slope estimate.
Time Frame: Predose on Days 1, 56, 154, and 182, 210 and at any time point on Days 14, 98, 189, 196, 203, and 238
Population: Population PK/PD analysis sample included all the participants with data available for PK/PD analysis.
Measure: Mean (90% Confidence Interval); unit: ms/[ng/mL]
Arm/Group | Delamanid
Number analyzed (Participants) | 37
ms/[ng/mL]
  Delamanid | 0.00792 [-0.00132 to 0.0172]
  Metabolite DM-6705 | 0.0613 [0.016 to 0.107]

12. Secondary Outcome: Number of Participants With Treatment Outcome as Assessed by Principal Investigator
Description: Treatment outcome was defined as favorable (cured and completed treatment) and unfavorable (lost to follow-up or died).
Time Frame: Month 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 12 to 17 Years of Age | Group 2: 6 to 11 Years of Age | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age
Number analyzed (Participants) | 7 | 6 | 12 | 12
Participants
  Favorable (Cured + Treatment Completed) | 6 | 6 | 10 | 11
  Unfavorable (Lost To Follow-up + Died) | 1 | 0 | 2 | 1

13. Secondary Outcome: Number of Participants With Abnormal Chest X-ray
Description: The data for the chest X-ray with abnormality, as assessed by investigator is reported.
Time Frame: From the first dose of study drug up to the end of the Post-treatment Follow-up Period (Up to Day 365)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 12 to 17 Years of Age | Group 2: 6 to 11 Years of Age | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age
Number analyzed (Participants) | 7 | 6 | 12 | 12
Participants | 7 | 6 | 12 | 11

14. Secondary Outcome: Number of Participants With Investigator-Assessed Signs and Symptoms of Tuberculosis
Description: The following signs and symptoms of tuberculosis were assessed by the investigator: cough, fever, weight loss, failure to thrive, hemoptysis, dyspnea, chest pain, night sweats and loss of appetite.
Time Frame: From the first dose of study drug up to the end of the Post-treatment Follow-up Period (Up to Day 365)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 12 to 17 Years of Age | Group 2: 6 to 11 Years of Age | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age
Number analyzed (Participants) | 7 | 6 | 12 | 12
Participants
  Cough | 6 | 4 | 3 | 7
  Fever | 1 | 2 | 2 | 5
  Weight Loss | 3 | 5 | 7 | 9
  Failure to Thrive | 0 | 1 | 0 | 3
  Hemoptysis | 2 | 0 | 0 | 0
  Dyspnea | 1 | 1 | 3 | 2
  Chest Pain | 1 | 1 | 0 | 0
  Night Sweats | 0 | 0 | 1 | 2
  Loss of Appetite | 1 | 2 | 2 | 6

15. Secondary Outcome: Sputum Culture Conversion (SCC)
Description: SCC was defined as a sputum specimen from a participant negative for growth of Mycobacterium tuberculosis (MTB), followed by at least one confirmatory negative sputum culture at least 27 days after the first negative sputum test and not followed by any sputum cultures positive for growth.
Time Frame: From the first dose of study drug up to the end of the Post-treatment Follow-up Period (Up to Day 365)
Population: Data for SCC could not be collected due to the paucity of sputum production in the participants.
Arm/Group | Group 1: 12 to 17 Years of Age | Group 2: 6 to 11 Years of Age | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Palatability Score as Assessed by the Investigator
Description: The palatability of the pediatric formulation was assessed using an age-appropriate visual hedonic scale and clinical assessment (Groups 3 and 4 only). The palatability result was based on 1 of 5 responses: 1=Dislike very much, 2=Dislike a little, 3=Neither liked nor disliked, 4=Like a little, 5=Like very much. Participants were categorized based on different scores. The data per the investigator score are reported.
Time Frame: Days 1, 28, 56 and 182
Population: Participants from the safety sample aged below 5 years (Groups 3 and 4) and who received any amount of IMP in this study, regardless of any protocol deviation or violation were analyzed for this outcome measure. Number analyzed is the number of participants with data available for analyses at the given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age
Number analyzed (Participants) | 12 | 12
Participants
  Day 1: Dislike Very Much | 0 | 0
  Day 1: Dislike a Little | 0 | 2
  Day 1: Neither Liked Nor Disliked | 1 | 0
  Day 1: Like a Little | 2 | 2
  Day 1: Like Very Much | 9 | 8
  Day 28: number analyzed (Participants) | 12 | 11
  Day 28: Dislike Very Much | 0 | 0
  Day 28: Dislike a Little | 0 | 0
  Day 28: Neither Liked Nor Disliked | 2 | 0
  Day 28: Like a Little | 1 | 2
  Day 28: Like Very Much | 9 | 9
  Day 56: number analyzed (Participants) | 12 | 11
  Day 56: Dislike Very Much | 0 | 0
  Day 56: Dislike a Little | 0 | 0
  Day 56: Neither Liked Nor Disliked | 0 | 0
  Day 56: Like a Little | 2 | 0
  Day 56: Like Very Much | 10 | 11
  Day 182: number analyzed (Participants) | 12 | 11
  Day 182: Dislike Very Much | 0 | 0
  Day 182: Dislike a Little | 0 | 1
  Day 182: Neither Liked Nor Disliked | 0 | 0
  Day 182: Like a Little | 1 | 5
  Day 182: Like Very Much | 11 | 5

17. Secondary Outcome: Number of Participants With Palatability Score as Assessed by the Parent or Participant
Description: The palatability of the pediatric formulation was assessed using an age-appropriate visual hedonic scale and clinical assessment (Groups 3 and 4 only). The palatability result was based on 1 of 5 responses: 1=Dislike very much, 2=Dislike a little, 3=Neither liked nor disliked, 4=Like a little, 5=Like very much. The data per parent/patient score are reported. Participants were categorized based on different scores.
Time Frame: Days 1, 28, 56 and 182
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age
Number analyzed (Participants) | 12 | 12
Participants
  Day 1: Dislike Very Much | 0 | 0
  Day 1: Dislike a Little | 0 | 1
  Day 1: Neither Liked Nor Disliked | 1 | 1
  Day 1: Like a Little | 2 | 3
  Day 1: Like Very Much | 9 | 7
  Day 28: number analyzed (Participants) | 12 | 11
  Day 28: Dislike Very Much | 0 | 0
  Day 28: Dislike a Little | 1 | 0
  Day 28: Neither Liked Nor Disliked | 0 | 0
  Day 28: Like a Little | 1 | 3
  Day 28: Like Very Much | 10 | 8
  Day 56: number analyzed (Participants) | 12 | 11
  Day 56: Dislike Very Much | 0 | 0
  Day 56: Dislike a Little | 0 | 0
  Day 56: Neither Liked Nor Disliked | 1 | 0
  Day 56: Like a Little | 0 | 0
  Day 56: Like Very Much | 11 | 11
  Day 182: number analyzed (Participants) | 12 | 11
  Day 182: Dislike Very Much | 0 | 0
  Day 182: Dislike a Little | 0 | 0
  Day 182: Neither Liked Nor Disliked | 0 | 1
  Day 182: Like a Little | 1 | 4
  Day 182: Like Very Much | 11 | 6

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to the end of the Post-treatment Follow-up Period (Up to Day 365)
Description: The Safety Sample included participants who received any amount of IMP in this study, regardless of any protocol deviation or violation.
Groups:
- Group 1: 12 to 17 Years of Age: Participants 12-17 years old (inclusive) received adult formulation of delamanid 100 mg (2x50 mg tablets), orally, BID plus OBR up to Day 182. Participants continued to receive OBR up to Day 365.
- Group 2: 6 to 11 Years of Age: Participants 6-11 years old (inclusive) received adult formulation delamanid 50 mg (1x50 mg tablet), orally, BID plus OBR up to Day 182. Participants continued to receive OBR up to Day 365.
Arm/Group | Group 1: 12 to 17 Years of Age | Group 2: 6 to 11 Years of Age | Group 3: 3 to 5 Years of Age | Group 4: Birth to 2 Years of Age
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 1/12 | 1/12
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/6 | 2/12 | 5/12
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 12/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 12 to 17 Years of Age (N=7) | Group 2: 6 to 11 Years of Age (N=6) | Group 3: 3 to 5 Years of Age (N=12) | Group 4: Birth to 2 Years of Age (N=12)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 12 to 17 Years of Age (N=7) | Group 2: 6 to 11 Years of Age (N=6) | Group 3: 3 to 5 Years of Age (N=12) | Group 4: Birth to 2 Years of Age (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Conductive deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 2 | 2
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 1
Vernal keratoconjunctivitis (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 2 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 3
Ascariasis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 1 | 4
Genital candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0
Helminthic infection (Infections and infestations) | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 2
Mumps (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 3
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0
Parasitic gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 2
Pharyngotonsillitis (Infections and infestations) | 1 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 3 | 2
Pustule (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0
Pyuria (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 4
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 2 | 0 | 0
Rubella (Infections and infestations) | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1
Systemic viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 5 | 2
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1
Tooth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood corticotrophin increased (Investigations) | 0 | 0 | 2 | 1
Coagulation time prolonged (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 2 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 2
Weight decreased (Investigations) | 0 | 0 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1 | 4 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Pain In extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 3 | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Sexual abuse (Social circumstances) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT01859923/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT01859923/SAP_001.pdf